CLINICAL TRIAL: NCT00922571
Title: A Study of Cataract Surgery With the Assistance of the Femtosecond Laser
Brief Title: A Study of Cataract Surgery With the Femtosecond Laser
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided not to pursue market release of prototype device used in this study
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OMC-C-1.1
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cataract
Keywords: Cataract; Femtosecond laser
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FS Laser Surgery (Experimental): For femtosecond laser-assisted cataract surgery (FS Laser Surgery), subjects will receive capsulotomy, lens segmentation and, at investigator discretion, lens softening using the OptiMedica Catalys™ Precision Laser System (Catalys System)
  Interventions: Procedure: FS Laser Surgery; Device: FS Laser System

INTERVENTIONS:
Procedure: FS Laser Surgery — The Catalys System is an ophthalmic surgical laser system intended for use in cataract surgery. The intervention consists of the both surgery and the use of the device.
Device: FS Laser System — The Catalys System is an ophthalmic surgical laser system intended for use in cataract surgery. The intervention consists of the both surgery and the use of the device.
  Other Names: OptiMedica Catalys™ Precision Laser System (Catalys System)

SUMMARY:
The purpose of this study is to evaluate the feasibility of using the Femtosecond Laser System to perform surgical maneuvers during cataract extraction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with the treatment/follow-up schedule and requirements
* Able to understand and provide written Informed Consent
* 3. ETDRS visual acuity equal to or worse than 20/30 (best corrected)
* Patient age between 50 and 80 years old
* Pupil dilates to at least 8 mm
* Patient able to fixate
* 1-3+ nuclear sclerotic cataract(This criterion does not apply to subjects who will receive post-IOL corneal relaxing incisions)
* Axial length between 22 and 26 mm

Exclusion Criteria:

* Pregnant, intending to become pregnant during course of study, less than 3 months postpartum or less than 6 weeks after completion of breast feeding
* Participation in a study of another device or drug within 3 months prior to study enrollment or during this study, and as per the Investigator's careful discretion, as long as not contradictory to any of the above criteria
* Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or for the study personnel) to treat the subject as part of this research study
* Anterior chamber depth less than 2.5 mm via Optical Coherence Tomography (Visante, Zeiss) or IOL Master (Zeiss) measurements
* History of prior ocular surgery
* History of ocular trauma
* Co-existing ocular disease affecting vision
* Astigmatism greater than five diopters (D.)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Capsulotomy Size | Day of Surgery
  Capsulotomy size will be measured during surgery.

SECONDARY OUTCOMES:
Cumulated Dissipated Energy (CDE) | Day of surgery
  CDE (the amount of ultrasound energy delivered during phacoemulsification of the crystalline lens) used will be measured during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Batlle, MD, Principal Investigator — Laser Center, Santo Domingo, Dominican Republic